CLINICAL TRIAL: NCT05480670
Title: Effect of Berberine Supplementation on Metabolic and Hormonal Features in Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Treatment Benefits of Berberine Supplementation for Women With PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayub Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ref. No. RC-2022/EA-01/178
Record Dates: First submitted 2022-07-24; First posted 2022-07-29 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Berberine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine arm (Experimental): Participants in this group will receive an oral 550 mg Berberine supplement tablet BDS for 3-months as an add-on to the changes in the diet/life-style for 3-months. The changes in the diet/life-style include limiting fat and carbohydrate intake and improve dietary behavior without the application of a calorie-restricted diet program. Exercise will also be recommended to include 30 min/day of moderate to intense activity.
  Interventions: Dietary Supplement: Berberine
- Control arm (No Intervention): Participants in this group will undergo changes in their diet/life-style.

INTERVENTIONS:
Dietary Supplement: Berberine — 550 mg Berberine supplement BDS for 3-months + changes in diet/life style.
  Arms: Berberine arm

SUMMARY:
Berberine is a plant alkaloid, reportedly possesses a wide range of pharmacological activities, including anti-obesity and anti-dyslipidemia. Berberine is an effective insulin sensitizer and has a comparable activity to MET in reducing IR. A large body of evidence suggest that Berberine dietary supplementation helps in improvement of symptoms associated with Polycystic Ovary Syndrome (PCOS). The purpose of this study is to investigate the treatment benefits of Berberine in women with PCOS.

DETAILED DESCRIPTION:
Berberine (BBR) is an isoquinoline derivative alkaloid that occurs in several plants including Oregon grape, barberry, tree turmeric, goldenseal, yellowroot, Amur corktree, Chinese goldthread, prickly poppy and Californian poppy.

Berberine supplementation has been suggested to improve the symptoms associated with PCOS. Berberine;

Reduces Insulin Resistance Lowers Blood Sugar Levels Aids in Weight Loss Improves Cholesterol Levels Regulates Menstrual Cycles Reduces Inflammation Helps Restore Hormonal Balance Improves Fertility Helps Combat Depression Helps Fight Fatty Liver Disease Improves Body Composition

The present RCT is aimed to investigate the effect of Berberine on these symptoms associated with PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 18 and 45 years
2. PCOS diagnosis as per the Rotterdam Criteria (any two of the following features:

   * Irregular periods (allso called oligomenorrea) or no periods (amenorrhea),
   * Higher levels of andregens present in the blood (hyperandrogenism), or physical characteristics of elevated andregen levels such as acne, male-pattern balding, or excess hair growth on face, chin, or body
   * Polycystic ovaries visible on an ultrasound
3. Normal, over-weight, and obese class I women (BMI 18.5 - 29.9 kg/m2, BMI cut-off as per the Asian criteria)
4. With no desire for pregnancy within 6 months
5. Able to give informed written consent

Exclusion Criteria:

1. Women who are currently taking or have teken in the last three months medications known to alter insulin physiology, oral contraceptives, ovulation induction drugs, anti- obesity or cholestrol lowering drugs, or any supplement known to interfere with insulin and androgen metabolism such as inositols, curcumin, lipoic acid, cinnamon, gymnemic and other botanical extracts.
2. Women undergoing in vitro fertilization treatment.
3. Women diagnosed with lateonset congenital adrenal hyperplasia (17-OH progestrone), thyroid disorders, hyperprolactinemia, diabetes mellitus and ODST.
4. Presence of liver, or renal disease
5. Pregnant or lactating or menopause women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Effect of Berberine on fasting blood glucose | up to 3 months
Effect of Berberine on fasting blood insulin | up to 3 months

SECONDARY OUTCOMES:
Effect of Berberine on physical sign and symptoms associated with PCOS | up to 3 months
  Effect on Hirsutism
Effect of Berberine on physical sign and symptoms associated with PCOS | up to 3 months
  Effect on Acne
Effect of Berberine on hormonal profile | up to 3 months
  Total testosterone
Effect of Berberine on hormonal profile | up to 3 months
  Sex hormone-binding globulin (SHBG)
Effect of Berberine on hormonal profile | up to 3 months
  Follicle stimulating hormone (FSH)
Effect of Berberine on hormonal profile | up to 3 months
  Luteinizing hormone (LH)
Effect of Berberine on hormonal profile | up to 3 months
  Anti-Mullerian hormone (AMH)
Effect of Berberine on fasting lipid metabolic profile | up to 3 months
  Total cholesterol
Effect of Berberine on fasting lipid metabolic profile | up to 3 months
  Total triglycerides (TG)
Effect of Berberine on fasting lipid metabolic profile | up to 3 months
  High density lipoprotein cholesterol (HDL-C)
Effect of Berberine on fasting lipid metabolic profile | up to 3 months
  Low density lipoprotein cholesterol (LDL-C)
Effect of Berberine on non-invasive markers of liver injury | up to 3 months
  ALT
Effect of Berberine on non-invasive markers of liver injury | up to 3 months
  AST
Effect of Berberine on non-invasive markers of liver injury | up to 3 months
  Gamma GT
Effect of Berberine on non-invasive markers of liver injury | up to 3 months
  Bilirubin
Effect of Berberine on non-invasive markers of liver injury | up to 3 months
  Alkaline phosphatase (ALP)

CONTACTS AND LOCATIONS:
Locations (1):
- Ayub Teaching Hospital, Abbottabad, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Pierro F, Sultana R, Eusaph AZ, Abrar S, Bugti M, Afridi F, Farooq U, Iqtadar S, Ghauri F, Makhduma S, Nourin S, Kanwal A, Bano A, Bugti AA, Mureed S, Ghazal A, Irshad R, Recchia M, Bertuccioli A, Putignano P, Riva A, Guasti L, Zerbinati N, Khan A. Effect of Berberine Phytosome on reproductive, dermatologic, and metabolic characteristics in women with polycystic ovary syndrome: a controlled, randomized, multi-centric, open-label clinical trial. Front Pharmacol. 2023 Nov 21;14:1269605. doi: 10.3389/fphar.2023.1269605. eCollection 2023. PMID 38074133